CLINICAL TRIAL: NCT07297485
Title: An Observational Cross-Sectional Comparison to Evaluate the Level of Agreement Between Standard Universal Goniometer Measurements and a Squat Height Calculator Algorithm to Determine Squat Position for Isometric Wall Squat Position.
Brief Title: Evaluating the Level of Agreement Between Goniometer Measurements and Algorithm to Determine Wall Squat Position
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Other Study IDs: 10240
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Wall Squat Position
Keywords: Goniometer; Algorithm; Wall Squat; Level of Agreement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wall Squat Position: Participants will have femur and fibula length (cm) measurements taken and complete both protocols unshod.
  Protocol 1 - Goniometer Squat Position Protocol A universal standard long arm goniometer will be aligned for knee flexion and held in position using soft velcro straps. A spirit level will establish and maintain vertical alignment of the fibula during the protocol. Participants will assume a 5-stage wall squat position. At each squat stage measurements for squat heigh at width will be recorded.
  Protocol 2 - Squat Height Calculator Femur and fibula bone measurements will be entered into the squat height calculator algorithm to determine the the 5-stage squat measurements.
  Markers will be placed on a squat height ruler for the height and width at each stage. Participants will be asked to align the lateral malleolus and greater trochanter with the markers and the joint angle measured using a universal standard long arm goniometer for each stage.

SUMMARY:
The wall squat exercise has been used in several research studies to help lower blood pressure. However, setting up the correct squat position often involves using a joint angle-measuring tool called a goniometer to get the knee at exactly the right angle. To set up the wall squat using a goniometer, someone has to stand in position, hold still while their knee angle is measured and adjusted, and then measure how high they should squat. This takes time, can be uncomfortable, and can be difficult to hold steady. This can make it difficult to get accurate measurements, particularly for people who are not used to exercise.

Therefore, the purpose of this research is to explore if a squat height calculator (based on leg bone measurements) to work out the squat height agrees with goniometer measurements for specific knee joint angles.

DETAILED DESCRIPTION:
The isometric wall squat exercise has been used as an intervention in several research studies However, how the protocol is delivered can vary between researchers; for example, participants can be instructed to adjust their foot position to keep lower leg vertical with the wall while lowering onto a squat position; while others use a standard goniometer in conjunction with a spirit level to establish knee joint angle and limb position. Therefore, to ensure study reliability and repeatability a standardised protocol to ensure consistent limb position needs to be established. Traditionally, measurement of joint angles and limb range of movement (ROM) using a standard universal goniometer is deemed gold standard in clinical settings. While the goniometer is portable and relatively inexpensive it has several limitations in terms of practical use. Firstly, both hands are required to align and stabilise the goniometer positioning, and maintaining the alignment during movement can be problematic. Also, the use of a standard universal goniometer requires alignment with specified bony landmarks, some of which are not visually located or palpated with ease and require a good level of underpinning anatomical knowledge. Moreover, the level of accuracy in goniometer alignment can be further reduced when observing intertester measurements. Consequently, challenges with goniometer alignment and stabilisation, alongside intertester variability, may lead to errors in measurement.

Using a standard universal goniometer in combination with a spirit level to establish the isometric wall squat position requires a baseline weight bearing position to be maintained while correct limb positions and knee joint angle are established, and squat height measurements recorded. This may be time consuming, uncomfortable, and difficult to maintain for untrained populations, particularly within the more acute degree angles, leading to difficulties in determining accurate baseline measurements. Therefore, an alternative method to determine squat position would be beneficial for the development and standardisation of the protocol. As linear bone growth typically ceases at ~18 yrs for females, and ~21yrs for males, limb length in the healthy adult population remains relatively consistent. Recent research has explored the use of artificial intelligence algorithms to predict overall height from femoral and tibial bone lengths. Therefore, based on this principle, this study aims to explore if using a squat height calculator algorithm, utilising lower limb bone lengths, agrees with gold standard universal goniometer measurements to ascertain positioning for an isometric wall squat at specific knee joint angles

ELIGIBILITY:
Inclusion Criteria:

* >21 years
* Written informed consent provided

Exclusion Criteria:

* Orthopaedic problems or injury affecting the hip, knee, or ankle joints
* Inability to stand unaided and hold a static position for >5 minutes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample recruited from the Tyne and Wear area.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Level of agreement | Baseline
  Level of agreement between standard long arm goniometer and squat height calculator algorithm will be determined at each squat stage for knee joint angle (degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Cucato, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon S, Fischer B, Rinner A, Hummer A, Frank BJH, Mitterer JA, Huber S, Aichmair A, Schwarz GM, Hofstaetter JG. Body height estimation from automated length measurements on standing long leg radiographs using artificial intelligence. Sci Rep. 2023 May 25;13(1):8504. doi: 10.1038/s41598-023-34670-2. PMID 37231033
- [Background] Kiatkulanusorn S, Luangpon N, Srijunto W, Watechagit S, Pitchayadejanant K, Kuharat S, Beg OA, Suato BP. Analysis of the concurrent validity and reliability of five common clinical goniometric devices. Sci Rep. 2023 Nov 27;13(1):20931. doi: 10.1038/s41598-023-48344-6. PMID 38017058
- [Background] Hanks J, Myers B. Validity, Reliability, and Efficiency of a Standard Goniometer, Medical Inclinometer, and Builder's Inclinometer. Int J Sports Phys Ther. 2023 Aug 1;18(4):989-996. doi: 10.26603/001c.83944. eCollection 2023. PMID 37547826
- [Background] Lea JWD, O'Driscoll JM, Hulbert S, Scales J, Wiles JD. Convergent Validity of Ratings of Perceived Exertion During Resistance Exercise in Healthy Participants: A Systematic Review and Meta-Analysis. Sports Med Open. 2022 Jan 8;8(1):2. doi: 10.1186/s40798-021-00386-8. PMID 35000021
- [Background] Wiles J, Rees-Roberts M, O'Driscoll JM, Doulton T, MacInnes D, Short V, Pellatt-Higgins T, Saxby K, Gousia K, West A, Smith M, Santer E, Darby J, Farmer CK. Feasibility study to assess the delivery of a novel isometric exercise intervention for people with stage 1 hypertension in the NHS: protocol for the IsoFIT-BP study including amendments to mitigate the risk of COVID-19. Pilot Feasibility Stud. 2021 Oct 28;7(1):192. doi: 10.1186/s40814-021-00925-w. PMID 34711266
- [Background] Lea JWD, O'Driscoll JM, Wiles JD. The implementation of a home-based isometric wall squat intervention using ratings of perceived exertion to select and control exercise intensity: a pilot study in normotensive and pre-hypertensive adults. Eur J Appl Physiol. 2024 Jan;124(1):281-293. doi: 10.1007/s00421-023-05269-2. Epub 2023 Jul 17. PMID 37458822